CLINICAL TRIAL: NCT07173556
Title: Evaluation of Safety, Tolerability, Efficacy, and Pharmacokinetic Characteristics of QLC1401 Tablets Combined With CDK4/6 Inhibitors or mTOR Inhibitors in Patients With Estrogen Receptor-Positive (ER+), Human Epidermal Growth Factor Receptor 2-Negative (HER2-) Locally Advanced or Metastatic Breast Cancer: A Phase Ib/II Clinical Study
Brief Title: A Phase Ib/II Study of QLC1401 Combined With CDK4/6 or mTOR Inhibitors in ER+/HER2- Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLC1401-201
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLC1401 in combination with CDK4/6 inhibitors (Experimental)
  Interventions: Drug: QLC1401
- QLC1401 in combination with mTOR inhibitors (Experimental)
  Interventions: Drug: QLC1401

INTERVENTIONS:
Drug: QLC1401 — CDK4/6 inhibitors: Palbociclib, Abemaciclib, Ribociclib
  Arms: QLC1401 in combination with CDK4/6 inhibitors
Drug: QLC1401 — mTOR inhibitors: Everolimus
  Arms: QLC1401 in combination with mTOR inhibitors

SUMMARY:
This study is an open-label, multicenter, Phase Ib/II clinical trial designed to evaluate the safety, tolerability, efficacy, and pharmacokinetic characteristics of QLC1401 tablets in combination with CDK4/6 inhibitors or mTOR inhibitors in patients with ER+/HER2- locally advanced or metastatic breast cancer. The study consists of two stages: a Phase Ib dose-escalation stage and a Phase II dose-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical trial, understand and sign the informed consent form, and agree to comply with the requirements specified in the protocol.
* Age ≥ 18 years.
* Female subjects must be postmenopausal and meet the trial requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* Life expectancy ≥ 3 months.
* Histologically or cytologically confirmed breast cancer.
* Based on the most recent biopsy results of primary or metastatic tumor tissue, immunohistochemistry (IHC) confirms ER-positive status and HER-2-negative status.
* At least one measurable target lesion according to RECIST v1.1.
* Adequate bone marrow function within 2 weeks (14 days) prior to the initiation of study treatment, without the need for transfusion or growth factor (G-CSF, EPO, TPO, etc.) support.
* Adequate liver function.
* Renal function: serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (Ccr) > 30 mL/min, with no significant electrolyte imbalances that are difficult to correct.
* Coagulation function: International Normalized Ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

Exclusion Criteria:

* Presence of symptomatic visceral disease or any other condition deemed unsuitable for endocrine therapy as per the investigator's judgment.
* Presence of unresolved toxicities from prior therapy that have not recovered to ≤ CTCAE grade 1, excluding alopecia (any grade) or other toxicities considered by the investigator to pose no safety risk.
* Received anti-tumor drug therapy within the specified time window prior to the first dose of the investigational drug.
* Prior treatment with an experimental SERD or experimental ER antagonist.
* Received radiotherapy within 4 weeks prior to the first dose of the investigational drug.
* Used a strong CYP3A4 inhibitor within 7 days or 5 half-lives (whichever is longer) prior to the first dose.
* Underwent major surgery within 4 weeks prior to the first dose of the investigational drug, or has not recovered from significant side effects, or has significant traumatic injury, non-healing wounds, or fractures.
* History of other active malignancies within 5 years prior to the first dose of the investigational drug.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Inability to swallow the formulation, or gastrointestinal impairment/disease that may affect adequate absorption of the investigational drug.
* Known clinically significant liver disease, including Child-Pugh class B or C, active viral hepatitis, or other hepatitis.
* Current documented grade 1 or higher pneumonitis or interstitial lung disease.
* Clinically significant pleural effusion, ascites, or pericardial effusion, defined as detectable on examination and requiring drainage within the past 2 weeks or additional medication to control symptoms.
* Clinically significant uncontrolled cardiac disease and/or recent cardiac events.
* History of bleeding tendency, thrombosis, or tumor embolism.
* Planned treatment with everolimus and presence of uncontrolled diabetes despite adequate therapy.
* Allergy to any of the investigational medicinal products or their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability (Phase Ib) | Throughout phase Ib (approximately 1 year)
  Types, incidence, and severity grades of AEs/SAEs and safety abnormalities, and their relationship to the investigational product; proportion of patients requiring dose adjustments or treatment discontinuation due to drug-related AEs.
Recommended phase II dose (RP2D) (Phase Ib) | Throughout phase Ib (approximately 1 year)
  RP2D will be selected upon safety, PK and efficacy data.
Objective Response Rate (ORR) (Phase II) | From time of Informed Consent to confirmed progressive disease (approximately 1 year)
  Objective Response Rate (ORR) as assessed by investigators per RECIST v1.1 criteria